CLINICAL TRIAL: NCT03281642
Title: Efficacy of a Nurse-based Intervention on Tobacco Consumption in Hospitalized Patients
Acronym: HOT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: HAO16020
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Smoking Patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Tobacco management — Training of healthcare teams for tobacco management by trained nurses. The intervention will consist of 3 minimum interviews, about 30 minutes each.
  Other Names: Training of healthcare teams for tobacco management

SUMMARY:
Tobacco consumption is a major public health problem, ranking second in the leading cause of morbidity and mortality worldwide, in 2010. The prevalence of tobacco smoking in hospitalized patients is evaluated around 20% and the management of tobacco reduction/cessation is an major issue for the course and outcome of many disorders.

Recent recommendations published by the French National Health Authority ("Haute Autorité de Santé", HAS) call for the involvement of all health professionals in helping patients to stop smoking and hospitalized patients are identified as a specific target. In addition, the meta-analysis of Rigotti et al. (2012) showed that the most effective programs (tobacco cessation) were those that include all patients, starting during the hospitalization with a specific follow-up of at least one month, and with the addition of nicotine replacement therapy. This combination increased the odds of successful tobacco cessation by 54%.

The project aims to evaluate the short-term efficacy (1 month) of a nurse-based program on tobacco smoking consumption in a population of hospitalized patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (>= 18 years), tobacco smokers, hospitalized in one of the participating unit during the inclusion period.
* For the sake of coherence with the literature, only subjects who smoked at least one cigarette a day in the previous 30 days before the hospitalization will be considered as "smokers".
* Affiliated to the national health system
* Signed informed consent

Exclusion Criteria:

* Patients enrolled in an addiction treatment during their hospitalization stay
* Cognitive deficit that makes the informed consent and the telephone interview impossible
* Aphasia
* Patient who does not speak French
* Life expectancy below 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All smoking patients hospitalized in one of the participating unit of the Saint-Louis-Lariboisière-Fernand Widal hospital (Diabetology, Cardiology, adults and adolescents Onco-hématology, Orthopedy, Oncology, Internal Medecine, Pneumology, Dermatology, Rhumatology, Psychiatry, Gastro-Entérology, Neurology) during the study period that include the 6 months preceding and the 6 months following the training.
Sampling Method: Non-Probability Sample
Enrollment: 430 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
1 month tobacco smoking prevalence | 1 month

SECONDARY OUTCOMES:
6 month tobacco smoking prevalence | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fernand Widal hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided